CLINICAL TRIAL: NCT01013948
Title: Prevalence of Chronic Airway Onstruction in a Subject Population With a History of Cigarette Smoking in a Primary Care Setting
Brief Title: Prevalence of Chronic Airway Obstruction in Subjects With a History of Cigarette Smoking in a Primary Care Setting
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111116
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Spirometry; Bronchitis; COPD; Chronic Obstructive Pulmonary Disease (COPD); Emphysema; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- N/A (Survey study)
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Investigational Product (Survey Study)

SUMMARY:
This is a cross-sectional study to determine the prevalence of symptomatic airway obstruction using the LFQ as a screening tool in primary care patients with a history of cigarette smoking and to provide descriptive data of this patient population. The study design is multicenter, cross-sectional, and involves a single visit. This study is not intended to evaluate the efficacy or safety of any investigational products. Following completion of written informed consent, eligible study subjects will complete a single study visit encompassing all required study assessments. Study subjects will not receive blinded study medication for evaluations of efficacy and safety.

All eligible patients will complete a self-administered Web survey that will include the LFQ. To meet both the primary and secondary aims, all patients with LFQ ≤ 18 (current cut-off for obstruction), as well as 5% of patients who score > 18, will be candidates for spirometric assessment. Only this subset of patients will undergo pulmonary function tests. Albuterol will be self-administered for determination of post-bronchodilator forced expiratory volume in one-second (FEV1)/forced vital capacity (FVC) ratio and post-bronchodilator FEV1 percentage of predicted normal. The study will end when 800 patients have been assessed spirometrically or 3,000 patients have completed the LFQ (whichever criterion is achieved first).

Prior to implementation of the full study, a pilot study will be conducted at two of the chosen study sites to pretest the proposed study procedures.

DETAILED DESCRIPTION:
The incidence of COPD is increasing throughout the world, with the vast majority of patients with the disease remaining undiagnosed (Coultas et al., 2001) and underreported (Frank et al., 2006; Global Initiative for Chronic Obstructive Lung Disease [GOLD], 2003; Peña et al., 2000; Takahashi et al., 2003; Van Weel et al., 2002). This is highlighted in a recent study that found 63% of patients with a smoking history and spirometry-confirmed COPD had no mention of COPD in their medical records (Frank et al., 2006). These findings are indicative of a low awareness of the condition among patients with COPD (Stratelis et al., 2004).

The use of patient-completed questionnaires to assess smoking history and status, respiratory symptoms, and socioeconomic status is a reliable and valid method of screening for COPD diagnosis and severity (Bednarek et al., 2008). The range of conditions described as COPD has led to confusion about disease terminology and difficulty with diagnosis and communication, particularly in primary care (Fukuhara et al., 2005; Kesten and Chapman, 1993). Considering that approximately 80% of patients diagnosed with COPD are current and previous cigarette smokers, mass screening of these populations using office-based spirometry becomes an attractive option (Furguson et al., 2000). A questionnaire designed to capture patient answers specific to their disease condition could provide invaluable information, which, if it correlates adequately with spirometry, could markedly improve diagnosis and provide avenues for appropriate treatment decisions. There are data supporting the argument that the prevalence of physician-diagnosed COPD is much lower than the prevalence suggested by results of population-based spirometric surveys (Chapman, 2004; Fukuchi et al., 2004; Peña et al., 2000; Soriano et al., 2000). Evidently, the development of a practical and reliable tool could help bridge the gaps in diagnosis and disease awareness. Moreover, prevalence studies underscore the need to improve awareness of COPD among cigarette-smoking populations and to provide information that could potentially lead patients to seek treatment. Hence, there is a need to develop a screening questionnaire able to identify patients at risk of airflow obstruction, for further evaluation. The LFQ, developed for this purpose, consists of a series of questions pertaining to COPD risk factors and symptoms.

Specifically, this study will aim to identify patients at risk of airflow obstruction as identified by the LFQ, the results of which will be followed for confirmation through subsequent spirometry in a subset of subjects. The LFQ will be evaluated against the spirometry results comparatively. A minimum age limit of 30 years is selected for subject participation in this study for further validation of the LFQ and to ascertain the enrollment of an adequately representative subset of subjects who may be bronchitic or asymptomatic for COPD, for comparison purposes with subjects with COPD. The study of this subject population may increase the sensitivity of COPD diagnosis and potentially provide information that could improve disease awareness and, as a consequence, possibly lead to optimization of disease management in primary care.

This is a cross-sectional study to determine the prevalence of symptomatic airway obstruction using the LFQ as a screening tool in primary care patients with a history of cigarette smoking and to provide descriptive data of this patient population. The study design is multicenter, cross-sectional, and involves a single visit. This study is not intended to evaluate the efficacy or safety of any investigational products. Following completion of written informed consent, eligible study subjects will complete a single study visit encompassing all required study assessments. Study subjects will not receive blinded study medication for evaluations of efficacy and safety.

All eligible patients will complete a self-administered Web survey that will include the LFQ. To meet both the primary and secondary aims, all patients with LFQ ≤ 18 (current cut-off for obstruction), as well as 5% of patients who score > 18, will be candidates for spirometric assessment. Only this subset of patients will undergo pulmonary function tests. Albuterol will be self-administered for determination of post-bronchodilator forced expiratory volume in one-second (FEV1)/forced vital capacity (FVC) ratio and post-bronchodilator FEV1 percentage of predicted normal. The study will end when 800 patients have been assessed spirometrically or 3,000 patients have completed the LFQ (whichever criterion is achieved first).

Prior to implementation of the full study, a pilot study will be conducted at two of the chosen study sites to pretest the proposed study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30 years or older
* Current or previous cigarette smoker with a history of cigarette smoking of ≥ 10 pack-years: number of pack years = (number of cigarettes per day/20) × number of years smoked) (e.g., 10 pack-years is equal to 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years). Previous smokers are defined as those who stopped smoking at least 3 months prior to the study visit.
* Willing and able to provide written informed consent prior to study participation (on day of study visit).
* Able to read, write, and comprehend information in English.

Exclusion Criteria:

* Prior to enrollment, prospective subjects will be screened. A subject will be excluded from the study if he/she meets any of the following criteria:
* Regular use (i.e., prescribed for use on a daily basis) of the following respiratory medications within the 4 weeks prior to the study visit:

  * Ipratropium (Atrovent, ipratropium bromide)
  * Ipratropium/albuterol combinations (e.g., Combivent)
  * Tiotropium (Spiriva, tiotropium bromide)
  * Salmeterol (SEREVENT™)
  * Formoterol (Foradil)
  * Inhaled corticosteroids (e.g., FLOVENT™, BECLOVENT™, Azmacort Aerobid, Pulmicort, QVAR, Vanceril)
  * Inhaled corticosteroid/long-acting beta-agonist combinations (e.g., ADVAIR DISKUS™ , Symbicort)
  * Theophyllines (e.g., Theo-dur, Slo-Bid, Uniphyl)
  * Oral beta-agonists (e.g.,Volmax)
* Previous lung surgery, including lung transplant, lung resection, lung volume reduction surgery (e.g., lobectomy, pneumonectomy).
* A known diagnosis of a significant lung condition including lung cancer, cystic fibrosis, pulmonary fibrosis, active tuberculosis, or sarcoidosis. A previous diagnosis of an obstructive lung disease is not exclusionary-asthma, chronic bronchitis, emphysema, alpha1-antitrypsin (A1AT) deficiency, etc.
* Current participation in a respiratory-related research study and receiving experimental medications.
* Limited ability to provide a valid informed consent due to serious uncontrolled psychiatric disease, intellectual or cognitive deficiency, poor motivation, current substance abuse (including drugs and alcohol), or other relevant condition that, in the opinion of the site principal investigator, will interfere with the subject's participation in the study.
* Pregnant females.
* Any medical or physical condition such as acute respiratory infection that would interfere with the adequate performance of spirometry.
* Participating investigator, sub-investigator, study coordinator, employee of the participating investigator, or family member of the aforementioned site staffs.

Ages: 30 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Current or previous cigarette smokers of at least 30 years of age with a history of cigarette smoking of ≥ 10 pack-years, recruited from primary care centers.
Sampling Method: Probability Sample
Enrollment: 1574 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome for this study will be the proportion of subjects at risk for airway obstruction as measured by the LFQ (LFQ total score ≤ 18) and confirmed by spirometry. | 4-Month

SECONDARY OUTCOMES:
Screening accuracy (sensitivity and specificity) of the LFQ utilizing spirometrically-defined airway obstruction (i.e., a post-bronchodilator FEV1/FVC ≤ 0.7). Proportion of patients with chronic airway obstruction as measured by the LFQ, stratified... | 4-Month

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (40):
  - GSK Investigational Site, Adamsville, Alabama
  - GSK Investigational Site, Foothill Ranch, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Los Gatos, California
  - GSK Investigational Site, Rolling Hills Estate, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Solana Beach, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Torrance/California, California
  - GSK Investigational Site, Tulare, California
  - GSK Investigational Site, Altmonte Springs, Florida
  - GSK Investigational Site, Belle Glade, Florida
  - GSK Investigational Site, Green Cove Springs, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Oviedo, Florida
  - GSK Investigational Site, Sebastian, Florida
  - GSK Investigational Site, Conyers, Georgia
  - GSK Investigational Site, Snellville, Georgia
  - GSK Investigational Site, Northbrook, Illinois
  - GSK Investigational Site, Vernon Hills, Illinois
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Williamsburg, Kentucky
  - GSK Investigational Site, Reisterstown, Maryland
  - GSK Investigational Site, West Plains, Missouri
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, Elmhurst, New York
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Cortland, Ohio
  - GSK Investigational Site, Lansdowne, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Flower Mound, Texas
  - GSK Investigational Site, Grand Prairie, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Richardson, Texas

REFERENCES:
- [Background] Mintz ML, Yawn BP, Mannino DM, Donohue JF, Hanania NA, Grellet CA, Gilsenan AW, McLeod LD, Dalal AA, Raphiou IH, Prillaman BA, Crater GD, Cicale MJ, Mapel DW. Prevalence of airway obstruction assessed by lung function questionnaire. Mayo Clin Proc. 2011 May;86(5):375-81. doi: 10.4065/mcp.2010.0787. PMID 21531880
- [Derived] Hanania NA, Crater GD, Morris AN, Emmett AH, O'Dell DM, Niewoehner DE. Benefits of adding fluticasone propionate/salmeterol to tiotropium in moderate to severe COPD. Respir Med. 2012 Jan;106(1):91-101. doi: 10.1016/j.rmed.2011.09.002. Epub 2011 Oct 29. PMID 22040533